CLINICAL TRIAL: NCT06483022
Title: Building Equitable Linkages With Interprofessional Education Valuing Everyone
Acronym: BELIEVE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-1258
Record Dates: First submitted 2024-06-13; First posted 2024-07-01 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Pregnancy Related; Postpartum; Pain
Keywords: Maternity Hospitals
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The investigators plan a multisite step-wedge cluster randomized trial to test the extent to which interprofessional collaboration training (IPC training) reduces racial disparities in postpartum pain (primary outcome) and pain assessment and treatment (secondary, health team processes), improves birthing people's experience of respectful care (secondary outcomes), and fostering a positive shift in health team interprofessional collaboration attitudes and teamwork (secondary process outcomes).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention (Placebo Comparator): In the pre-intervention sequence(s), birthing people at participating hospitals will experience treatment-as-usual.
  Interventions: Other: Usual Care
- Post-intervention (Active Comparator): In the post-intervention sequence(s), birthing people at participating hospitals will experience treatment by health care teams that have undergone the Building Equitable Linkages With Interprofessional Education Valuing Everyone interprofessional education (BELIEVE IPE) training.
  Interventions: Behavioral: BELIEVE IPE Training

INTERVENTIONS:
Behavioral: BELIEVE IPE Training — The IPC training will be delivered to health team members who provide intrapartum and/or postpartum maternity care at each facility. Individuals with roles as maternity care providers, nurses, lactation consultants or doulas whose primary inpatient clinical assignment is maternity care will be included in the training. The training will consist of a pre-session module (about 60 minutes), a 90-minute interprofessional collaboration session, delivered using virtual reality head-sets, and post-session modules (about 60 minutes). The pre- and post-session modules will be delivered through an online learning platform.
  Arms: Post-intervention
Other: Usual Care — Prior to implementation of the IPC training, birthing people at the facilities will receive treatment-as-usual
  Arms: Pre-intervention

SUMMARY:
This is a step-wedge design implementation protocol of an interprofessional education curriculum intervention that is delivered through virtual reality and designed to reduce disparities and improve patient experiences in receiving maternal healthcare.

ELIGIBILITY:
Inclusion Criteria:

Healthcare Team Participants

* Employed as one of the following roles: maternity care provider, nurse, lactation consultant or doula.
* Primary inpatient clinical assignment is maternity care.
* If Per Diem: Employed for a minimum of 4 shifts/month at a participating site.

Birthing Parent Data Extraction Participants

• Had a live birth at a participating site from the start of the study through the last Data Retrieval timepoint.

Birthing Parent Interview Participants

* Had a live birth at a participating site from the start of the study through the last Data Retrieval timepoint.
* Black race or Limited English Proficiency with preferred language of Spanish.
* Age ≥ 18.

Exclusion Criteria:

Healthcare Team Participants

• None

Birthing Parent Data Extraction Participants

• Baby with birth gestational age < 24 weeks.

Birthing Parent Interview Participants

* Baby with birth gestational age < 24 weeks.
* Baby is no longer alive at time of Data Retrieval (regardless of gestational age).
* Currently incarcerated.
* Previously completed a birthing parent interview for the BELIEVE study.
* Previously enrolled as a Healthcare Team Participant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32000 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Severe Postpartum Pain | 0 to <24 and 24 to <48 hours postpartum
  Proportion of individuals with severe pain postpartum. Severe pain will be defined as pain score >4 on postpartum day 1 following vaginal birth, or pain score >7 on postpartum day 2 following cesarean birth, as documented in the electronic health record using the Numerical Rating Scale (NRS) of patient-reported pain from 0-10.

SECONDARY OUTCOMES:
Birthing parent-reported experiences of the respectful care (Qualitative) | 2-8 weeks postpartum
  Based on semi-structured interviews with a subset of birthing parents, the investigators will report the count of qualitative interview participants who described their care as "respectful" during semi-structured interviews with birthing parents.
Patient-reported examples of respectful and equitable health care team member practices (Qualitative) | 2-8 weeks postpartum
  Based on semi-structured interviews with a subset of birthing parents, the investigators will identify respectful and equitable health care team member practices in a thematic coded content analysis of transcribed responses. For the top three practices identified, the count of participants naming each practice will be reported.
Patient-reported examples of supportive health team member practices for pain management (Qualitative) | 2-8 weeks postpartum
  Based on semi-structured interviews with a subset of birthing parents, the investigators will identify supportive health team member practices for pain management in a thematic coded content analysis of transcribed responses. For the top three practices identified, the count of participants naming each practice will be reported.
Pain assessments | 0 to <24 and 24 to <48 hours postpartum
  Number of instances of pain score assessments on a 0-10 scale that are documented in the birthing parent's medical record.
NSAID doses administered | 0 to <24 and 24 to <48 hours postpartum
  Number of non-steroidal anti-inflammatory (NSAID) doses administered to the birthing parent, as documented in the medication administration record (MAR).
MMEs administered | 0 to <24 and 24 to <48 hours postpartum
  Number of Morphine Milligram Equivalents (MMEs) of opioids administered to the birthing parent, as documented in the medication administration record (MAR).
Acetaminophen doses administered | 0 to <24 and 24 to <48 hours postpartum
  Number of Acetaminophen doses administered to the birthing parent, as documented in the medication administration record (MAR).
Healthcare team members' perceptions of interprofessional collaboration | Baseline (pre-intervention) and after completing the IPC training intervention, a total of up to 4 months
  Using the modified Interprofessional Attitudes Scale (IPAS), attitudes of health care team members toward collaboration will be assessed. The IPAS is a 5-point Likert scale with scores ranging from 27 to 135, with higher scores reflecting more positive attitudes toward interprofessional collaboration.
Quality of interprofessional teamwork | Baseline (pre-intervention) and after completing the IPC training intervention, a total of up to 4 months
  Utilizing the modified Assessment for Collaborative Environments (ACE) Scale, health care team member perceptions of interprofessional communication will be assessed. The modified ACE is a 4-point Likert scale with scores ranging from 6 to 24, with higher scores reflecting better quality interprofessional teamwork.
Feasibility of the IPC training | 2-8 weeks after health care team members' completion of the IPC training
  Based on semi-structured interviews collected post intervention among a subset of health care team members, the investigators will conduct thematic coded content analysis of transcribed responses. The investigators will report the count of health care team members who described the intervention as feasible. Feasibility is defined as a positive rating about the intervention's potential performance in real-life conditions in birthing hospitals.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Stuebe, MD, MSc, Principal Investigator — University of North Carollina at Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC and Cone Health.
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC or REB and an executed data use/sharing agreement with UNC and Cone Health.